CLINICAL TRIAL: NCT00932347
Title: Effect of Mouthwash Containing Camellia Sinensis Extracts on Oral Malodor, Plaque and Papillary Bleeding Indices in Gingivitis Patients.
Brief Title: Effect of Mouthwash Containing Camellia Sinensis Extracts on Oral Malodor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Supanee Rassameemasmaung, Department of Oral Medicine, Faculty of Dentistry, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COA. No. MU-IRB 2008/177.1211
Record Dates: First submitted 2009-07-01; First posted 2009-07-03 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-07

CONDITIONS: Gingivitis; Halitosis
Keywords: Camellia sinensis; volatile sulfur compounds
MeSH Terms: conditions — Gingivitis; Halitosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mouthwash A (Experimental): Mouthwash A: Camellia sinensis mouthwash
  Interventions: Drug: Camellia sinensis mouthwash
- Mouthwash B (Placebo Comparator): Mouthwash B: Placebo mouthwash
  Interventions: Drug: Placebo mouthwash

INTERVENTIONS:
Drug: Camellia sinensis mouthwash — mouthrinsing, 2 times/day, for 28 days
  Other Names: Green tea mouthwash
  Arms: Mouthwash A
Drug: Placebo mouthwash — mouthrinsing, 2 times/day, for 28 days
  Other Names: placebo
  Arms: Mouthwash B

SUMMARY:
The purpose of this study is to determine effect of Mouthwash containing Camellia sinensis extracts on oral malodor and gingival inflammation in gingivitis subjects.

DETAILED DESCRIPTION:
At baseline, level of volatile sulfur compounds (VSC) in mouth air, Plaque Index and Papillary Bleeding Index will be recorded. Gingivitis subjects will be asked to rinse with Camellia sinensis mouthwash or placebo mouthwash. VSC level will be measured at 30 minutes and 3 hours post-rinsing. For the following 4 weeks, subjects will be rinsed with the assigned mouthwash twice daily after toothbrushing. All parameter will be recorded again at Day 28.

ELIGIBILITY:
Inclusion Criteria:

* at least 20 teeth
* clinical diagnosis as plaque induced gingivitis
* having over 80 ppb of volatile sulfur compounds in mouth air

Exclusion Criteria:

* smoker
* denture wearer
* having systemic diseases or oral pathology
* taking antibiotics 1 month prior to study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-09 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
level of volatile sulfur compounds in mouth air (part per billion) | baseline, 30 minutes, 3 hours, 28 days

SECONDARY OUTCOMES:
Papillary bleeding index | baseline, 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Supanee Rassameemasmaung, Ph.D, Principal Investigator — Department of Oral Medicine, Faculty of Dentistry, Mahidol University
Locations (2):
- Thailand (2):
  - Post Graduate Clinic 2, Faculty of Dentistry, Mahidol University, Bangkok, Bangkok
  - Post Graduate Clinic 2, Faculty of Dentistry, Mahidol University, Bangkok